CLINICAL TRIAL: NCT00542334
Title: Prevalence of Nocturnal Hypoglycemia in Children and Adolescents With Type 1 Diabetes on a Standard (TID) Insulin Regimen Using a Continuous Glucose Monitoring System (CGMS) - A Pilot Study
Brief Title: Prevalence of Nocturnal Hypoglycemia in Children on a Type 1 Diabetes (TID) Insulin Regimen Using a Continuous Glucose Monitoring System (CGMS)
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Alexandra Ahmet, Principal Investigator- MD,BSc, FRCPC, Children's Hospital of Eastern Ontario
Other Study IDs: 07/02S(E)
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Nocturnal Hypoglycemia; Type 1 Diabetes
Keywords: Nocturnal Hypoglycemia; Type 1 diabetes; Children; Adolescents; CGMS
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will help determine the frequency and magnitude of nocturnal hypoglycemia (low blood sugar at night during sleep), in children with type 1 diabetes who are on a standard insulin regimen, by using a Continuous Glucose Monitoring System (CGMS). Secondary objectives include the establishment of a definition of nocturnal hypoglycemia for the CGMS and for the calculation of sample size needed for future studies using CGMS. Nocturnal hypoglycemia (NH) can be associated with significant morbidity including seizure and coma. The investigators intend to use the CGMS in a future study investigating the use of a new insulin combination aimed to decrease the frequency of NH in the pediatric population.

Thirty pediatric subjects with established type 1 diabetes mellitus will be asked to wear a CGMS for 3 days. During this time the participants will be required to test and record self-monitored blood glucose readings at designated time periods and if they have symptoms of hypoglycemia. The comparison of these values with each other and with different previously defined values of NH will allow for a clear definition of NH to be made. A survey has also been designed to assess participant satisfaction with the CGMS.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* less than 18 years of age
* >2 year duration of diabetes
* on a conventional TID insulin regimen (morning and bedtime NPH) for a minimum of 3 months
* informed consent and assent

Exclusion Criteria:

* medical conditions other than treated hypothyroidism or asthma requiring oral glucocorticoids more than once per year
* intention to move outside of CHEO's catchment area within the next 4 months
* more than 17 years of age and unwilling to continue receiving diabetes care at CHEO until study completion
* intention to switch to a different insulin regimen prior to study completion

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents with type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Frequency and magnitude of nocturnal hypoglycemia | 3 days

SECONDARY OUTCOMES:
Patient satisfaction with continuous glucose sensing | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra H Ahmet, MD, BSc,FRCPC, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hosiptal of Eastern Ontario, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Ahmet A, Dagenais S, Barrowman NJ, Collins CJ, Lawson ML. Prevalence of nocturnal hypoglycemia in pediatric type 1 diabetes: a pilot study using continuous glucose monitoring. J Pediatr. 2011 Aug;159(2):297-302.e1. doi: 10.1016/j.jpeds.2011.01.064. Epub 2011 Mar 17. PMID 21414634